CLINICAL TRIAL: NCT03457324
Title: Efficacy and Safety of Chinese Medicine JCM-16021 for Diarrhea-predominant Irritable Bowel Syndrome: a Multicenter, Randomized, Double-blind, Placebo Controlled Clinical Trial
Brief Title: Efficacy and Safety of Chinese Medicine JCM-16021 for Diarrhea-predominant Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhaoXiang Bian (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, ZhaoXiang Bian, Chair Professor of Clinical Division, Hong Kong Baptist University
Organization: Hong Kong Baptist University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITS-148-14FP
Record Dates: First submitted 2018-02-08; First posted 2018-03-07 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: JCM-16021; Trial; Irritable Bowel Syndrome; Chinese Medicine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — JCM-16021

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JCM-16021 Group (Experimental): JCM-16021 granules 8g/sachet, three times daily for 8 weeks.
  Interventions: Drug: JCM-16021
- Placebo Group (Placebo Comparator): Placebo granules 8g/sachet, three times daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JCM-16021 — This prescription with seven ingredients.
  Arms: JCM-16021 Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo controlled clinical trial, in order to evaluate the efficacy and safety of Chinese Medicine JCM-16021 for diarrhea-predominant irritable bowel syndrome. All patients will be evaluated for study eligibility at Visits 1 (baseline) and 2 (2 weeks). On visit 2, patients who meet the criteria will be randomly assigned to receive 8-week treatment of either JCM-16021 Granules or JCM-16021 placebo Granules. The investigators, research assistants and participants are not aware of the treatment assignments throughout the study. Treatment codes will only be broken after the completion of study. The assessments at Visit 3 (4-week post treatment) and at visit 4 (end of 8-week treatment) are used to measure treatment response (i.e. changes from baseline). Assessment at visit 5 (end of 8-week follow up) is to determine any sustained response to treatment. All the visits will be carried out in HKBU and CUHK clinics.

DETAILED DESCRIPTION:
Sample size calculation:

Sample size is calculated on the basis of primary efficacy variables. From our previous study, the global assessment of improvement (GAI) were 52% in herbal medicine group and 32% in western medicine group, respectively. According to the references (Corazziari E, Bytzer P, Delvaux M, et al. Clinical trial guidelines for pharmacological treatment of irritable bowel syndrome. Alimentary pharmacology & therapeutics 2003; 18 (6): 569-580), the investigational drug is more effective than placebo (the overall improvement rate of symptoms is 15%), using StudySize2.0 software to calculate the sample size, assuming the improvement in the treatment group is 52%. In order to detect a difference with a two-side p value <0.05 and 80% statistical power, we will need to recruit 166 patients per arm. Further assuming a 15% dropout rate, we conclude that a total of 392 patients (196 per arm) will be recruited to ensure statistically significant results.For the number of cases distribution between centers, according to the references (Lai D,Chang KC, Rahbar MH, Moye LA. Optimal Allocation of Sample Sizes to Multicenter Clinical Trials. Journal of biopharmaceutical statistics 2013; 23 (4): 818-828) , from the following equation, we will consider the center about the patient flow, traffic, treatment,costs and other possible factors, we will use the formula below to estimate the number of cases that will be recruited in each center.

Research medical record and Electronic Database:

All patients should be observed and assessed based on clinical trial protocol and the investigators need to document in the medical record accurately and clearly. Research medical record is the source document which cannot be altered. Any correction should not change the original record and can only be added in a way of narration with reasons. The doctor participated in the clinical trial needs to sign and date the record. An electronic database will be created. Each study site will input their own data and be responsible for its accuracy. A chief statistician will be responsible for data cleaning and data analysis.

Analysis parameters:

All parameters and study elements will be analyzed. The statistical analysis will be performed using SAS 9.1 and SPSS software.

Analysis sets:

Full analysis set (FAS): The analysis will be conducted according to the intention-to-treat (ITT) principle which means to eliminate the participants with a minimum and reasonable method. ITT population refers to all participants who go through randomization, enter double-blind treatment period, and receive IMP at least one time. Missing values of efficacy will be imputed by the last-observation-carried forward (LOCF) method. Per-protocol set (PP): PP population refers to all participants who complete relative observation according to protocol requirement and are confirmed to meet following conditions: ① compliance between 80% and 120%; ② not taking probihited medications during the process of trial; ③ meeting inclusion criteria and not fitting any exclusion items; ④ completing all planned visits and necessary items of CRF. Missing values of this set will still be processed as missing data and not be imputed. Safety analysis set: Population for safety analysis refers to all participants who enter the trial, receive medication at least one time and have suitable follow-up data for safety analysis. All safety data including AEs and laboratory results from participants will be assessed.16.3 Statistical analysis technique Baseline data (gender, age, race, weight, height, vital signs, course of IBS, history of smoking and alcohol) will be descriptively summarized. Differences of measurement data between the groups will be assessed with the use of t-test for normally distributed continuous variables and Wilcoxon signed rank test for non-normally distributed. Differences of enumeration data between the groups will be assessed with the use of chi-square test or CMH test when considering multicenter character. Measurement data of different groups in each visit will be reported as mean ± standard deviation (SD). Intra-group comparisons between baseline and each visit will be conducted by using paired t-test (or Wilcoxon signed rank test). Comparisons between groups will be conducted by using an analysis of variance (ANOVA), with other confounding factors like multicenter character conducting the covariate analysis. Statistical analysis for the data which do not meet above conditions (e.g. non-normal) will be conducted with the use of non-parametric test. Enumeration data of different groups in each visit will be reported as frequency (proportion). Comparisons between groups will be assessed with the use of X2 test (CMH test) or non-parametric test. Dropout analysis: Dropout analysis will be conducted with the use of chi-square test. If the data do not conform to chi-square test (data include 0, or theoretical frequency is below 1), Fisher's exact test will be used. Compliance analysis: Compliance analysis will be conducted with the use of chi-square test. If the data do not conform to chi-square test (data include 0, or theoretical frequency is below 1), Fisher's exact test will be used.

Hypothesis testing:

This trial will conduct superiority analysis firstly. Other difference test will be conduct by two-sided test. The statistical significance will be defined as two-sided P-value of ≤0.05 without any special explanation.

Efficacy analysis:

The efficacy analysis will be conducted with the use of PP analysis and ITT analysis in the meantime. Comparisons of measurement data will be conducted by using analysis of covariance (ANCOVA), with treatment group and trial center as a factor in the model and baseline as the covariate. Comparisons of measurement data will be conducted by using chi-square test or CMH chi-square test when considering multicenter character. Meanwhile, superiority analysis between experimental group and control group will be conducted based on primary efficacy variables. Superiority test depends on interval method.

Safety analysis:

Extent of exposure: Descriptive statistics will be conducted according to the exposure dose and time of medication in different groups. AEs analysis: Comparisons of incidence rate of AEs between groups will be conducted with the use of X2 test. And investigators need to list and describe the AEs happened in this trial. If the data do not conform to X2 test (data include 0, or theoretical frequency is below 5), Fisher's exact test will be used.

Data management:

CRFs are filled in by investigators and study coordinators, other assessment forms by every participant (including dropout cases). Data processing will be conducted in accordance with the following protocol:

1. Verification of CRFs: Study coordinators need to verify CRFs before inputting.
2. Data verification needs to be conducted successively in the following two steps:

   1. Verify the consistency and logicality of data: Review contents of data range and logicality are determined by the range of each indexes and the interrelation. Corresponding software will also be written to correct the incorrect data.
   2. Compare database and CRFs by manual testing. Selectively counter check 10% CRFs with participants' medical notes to know the quality of inputting and analyze and handle the existing problems.
3. Data inspection and closure of database: After verifying the validity of established database and statistical protocol, principal investigators, will lock the data. The locked data are not allowed to change. Confirmed problems found after locking will be handled in the process of statistical analysis. All mistakes and modification should be recorded and kept properly.

ELIGIBILITY:
Inclusion Criteria:

1. fulfill the diagnostic criteria of diarrhea-predominant IBS (IBS-D);
2. fulfill the diagnostic criteria of diarrhea with TCM pattern of liver depression and spleen deficiency (LDSD);
3. age of 18-65 years (inclusive);
4. participants are voluntary and provide written informed consent.

Exclusion Criteria:

1. constipation-predominant, mixed or unsubtyped IBS patients;
2. severe diseases on heart, liver and kidney, hematology or cancer which is diagnosed by traditional Chinese medicines;
3. medical history of organic gastrointestinal diseases (e.g. inflammatory bowel diseases, intestinal tuberculosis, colon polyps), or systemic diseases which could affect gastrointestinal motility (e.g. hyperthyroidism, diabetes mellitus, chronic renal failure, neuropsychiatric diseases) which is diagnosed by traditional Chinese medicines;
4. current concomitant medication with effects on gastrointestinal function (e.g. anticholinergic drugs, calcium channel blockers, 5-HT3 receptor antagonists, antidiarrheal agents, antacids, prokinetic agents, antidepressants, anxiolytics and intestinal flora regulating drugs);
5. medical history of abdominal surgery (e.g. cholecystectomy, etc.);
6. drug or food allergies;
7. pregnancy or breast-feeding;
8. medical history of neurological diseases or psychiatric disorders;
9. currently participating in another clinical trial;
10. taking IBS treatment drugs within 1 week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Global Assessment of Improvement (GAI) score | 16 weeks
  The global symptom improvement will be evaluated by scales (terrible=0, worse=1, slightly worse=2, no change=3, slightly better=4, better=5, excellent=6).

SECONDARY OUTCOMES:
Pain responder rate in daily worst abdominal pain scores | 16 weeks
  Pain responders are defined as that participants who met the daily pain response criteria for at least 50% of the days with diary entries during the observational period of interest. Daily pain response: decrease in the worst abdominal pain scores in the past 24 hours of ≥ 30% compared to baseline (average of daily worst abdominal pain the 2-week prior to randomization). Pain score is ranked from 0 to 10 represented none to most severe.
Stool consistency responder rate In daily stool consistency scores | 16 weeks
  Stool consistency responders are defined as that participants who met daily stool consistency response criterion (ie, score of 1, 2, 3, or 4 or absence of bowel movement if accompanied by ≥30% decrease in worst abdominal pain scores compared to baseline pain) for at least 50% of days with diary entries during the observational period of interest. Bristol stool scale is defined as 7-point Scale in which a score of 1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = sausage-like with cracks on the surface, 4 = sausage-like but smooth and soft, 5 = soft blobs with clear cut edges, 6 = fluffy pieces with ragged edges, and 7 = watery with no solid pieces.
Efficacy judgement standard of single symptom | 16 weeks
  1. Excellent: symptom disappearing;
  2. Effective: symptom decreased, scoring declining more than 2 points (including 2 points);
  3. Helpful: symptom decreased, scoring declining between 1 point to 2 points;
  4. Invalid: no change in symptom. Improvement contains excellent, effective and helpful. Each cardinal symptom total improvement rate will be calculated and then conducted symptom evaluation.
Comprehensive efficacy judgement standard of cardinal symptoms | 16 weeks
  The symptom improvement rate is calculated by "(total scoring of prior treatment - total scoring of post treatment) / total scoring of prior treatment × 100%". Clinical remission is defined as symptom disappearing, symptom improvement rate equal or greater than 80% is excellent, symptom improvement rate between 50% and 80% is helpful, symptom improvement rate under 50% is invalid, and negative symptom improvement rate is deterioration. Total effective rate is based on recovery and excellent cases.
TCM pattern improvement | 16 weeks
  Clinical remission: clinical symptoms and signs disappear or basically disappear, total scoring declining ≥95%; Excellence: clinical symptoms and signs are significantly improved, total scoring declining ≥ 70%; Effective: clinical symptoms and signs are improved, total scoring declining ≥ 30%; Invalid: clinical symptoms and signs are without obvious improvement or even with exacerbation, total scoring declining < 30%. Remark: calculation formula (nimodipine method) is: [(scoring of prior treatment - scoring of post treatment) / scoring of prior treatment]×100%
Quality of life scoring (IBS-QoL) | 16 weeks
  IBS-QoL includes 34 items and divides into 8 subscales, i.e. dysphoria (Q1), interference with activity (Q2), body image (Q3), health worry (Q4), food avoidance (Q5), social reaction (Q6), sexual (Q7) and relationship (Q8). Each item has a five-point response scale with reverse scoring. After conversion, total scoring will be in 0-100 range. Higher scoring reflects superior quality of life.
Irritable Bowel Syndromes-Symptom Severity Score (IBS-SSS) | 16 weeks
  The IBS-SSS is involved five aspects: the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal discomfort, defecation satisfaction, and interference with daily life. The range of score is 0-500 points scale.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Wu, M.D., Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Chinese Medicine Clinics of Hong Kong Baptist University, Hong Kong, Hong Kong
  - Institute of Digestive Disease, The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
We will submit the study protocol and clinical study report with the informed consent form for publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The study protocol will be submitted during study recruitment, while the clinical study report with the informed consent form will be submitted within 1 year after the completion of study.
Access Criteria: All researchers can get the information by sending requests to the study contact person.

REFERENCES:
- [Derived] Zhai L, Zheng Y, Lo CW, Xu S, Jiang X, Liu Q, Ching JY, Ning Z, Bao G, Yang W, Zhang Q, Cheng CW, Lam WC, Chan KL, Zhang X, Lam PY, Wu XY, Zhong LLD, Cao PH, Koh M, Cheong PK, Lin Z, Lin C, Zhao L, Wong XHL, Wu JC, Bian Z. Butyrate-producing commensal bacteria mediates the efficacy of herbal medicine JCM-16021 on abdominal pain in diarrhea-predominant irritable bowel syndrome: a randomized clinical trial. Phytomedicine. 2025 Sep;145:157040. doi: 10.1016/j.phymed.2025.157040. Epub 2025 Jul 1. PMID 40639240
- [Derived] Zheng Y, Ching J, Cheng CW, Lam WC, Chan KL, Zhang X, Lam PY, Wu XY, Zhong LLD, Cao PH, Lo CW, Cheong PK, Lin Z, Koh M, Wu J, Bian ZX. Efficacy and safety of Chinese medicine JCM-16021 for diarrhea-predominant irritable bowel syndrome: study protocol for a multi-center, randomized, double-blind, placebo controlled clinical trial. Chin Med. 2021 Nov 13;16(1):117. doi: 10.1186/s13020-021-00530-2. PMID 34774080